CLINICAL TRIAL: NCT06821308
Title: A Randomized Controlled Clinical Trial to Assess Crestal Bone Remodeling of Four Different Implant Designs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC/2015/0338/AM02
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2015-06

CONDITIONS: Dental Implant Bone Loss
Keywords: Dental implant, crestal bone loss, microthreads, implant-abutment connection

STUDY DESIGN:
Intervention Model Description: Split-mouth study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Internal Microthread implant (Active Comparator): Each participant received 4 implants, one of each type
  Interventions: Device: Implant placement
- Internal Non Microthread implant (Experimental)
  Interventions: Device: Implant placement
- External microthread implant (Experimental)
  Interventions: Device: Implant placement
- External Non-Microthread implant (Experimental)
  Interventions: Device: Implant placement

INTERVENTIONS:
Device: Implant placement — Each patient received 4 implants to support a bar supported overdenture. One implant is commercially available, 3 implants were experimentally made by the manufacturer for this study. The implants were similar in macro-desing, surface and platform shift but differ in microthread design and implant-abutment connection.

SUMMARY:
This randomized controlled trial aimed to assess the effect of the implant neck design (microthreaded vs. non-microthreaded) as well as the type of abutment connection (internal conical vs. external flat-to-flat) on long-term crestal bone remodelling and peri-implant health. Four implants used for a bar-retained maxillary overdenture, were followed over a period of at least 6 years.

Twenty-five patients were treated with a bar-retained maxillary overdenture. Four different implants were placed, with respectively: internal connection and microthreads on the implant neck (I MT); internal connection, without microthreads (I NMT); external connection, with microthreads (E MT); and external connection, without microthreads (E NMT). Other design features, s.a. diameter, surface topography, extent of platform switch as well as the surgical and prosthetic treatment protocol were identical. Radiographic crestal bone loss (CBL), plaque score (PS), bleeding on probing (Bop) and probing pocket depth (PPD) were determined at 1 and 6 years after implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Edentulous in the maxilla and sufficient bone to harvest four 4 x 9 mm implant

Exclusion Criteria:

* Head -and neck radiation
* Bisphosphonate intake
* Limited prosthetic height

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09-18 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Crestal bone loss | The measurements were performed at 1 and 6 years
  Radiographic measurement of crestal bone loss

SECONDARY OUTCOMES:
Plaque | The measurements were performed at 1 and 6 years
  Plaque was measured at 4 sites on each implant
Probing pocket depth | The measurements were performed at 1 and 6 years
Bleeding on probing | The measurements were performed at 1 and 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Hugo De Bruyn, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doornewaard R, Sakani S, Matthys C, Glibert M, Bronkhorst E, Vandeweghe S, Vervaeke S, De Bruyn H. Four-implant-supported overdenture treatment in the maxilla. Part I: A randomized controlled split mouth trial assessing the effect of microthreads and abutment connection type on 4 years peri-implant health. Clin Implant Dent Relat Res. 2021 Oct;23(5):671-679. doi: 10.1111/cid.13037. Epub 2021 Aug 11. PMID 34378860
- [Background] Glibert M, Vervaeke S, Jacquet W, Vermeersch K, Ostman PO, De Bruyn H. A randomized controlled clinical trial to assess crestal bone remodeling of four different implant designs. Clin Implant Dent Relat Res. 2018 Aug;20(4):455-462. doi: 10.1111/cid.12604. Epub 2018 Mar 25. PMID 29575488
- [Derived] Matthijs S, Christiaens V, Matthys C, De Bruyn H, Glibert M. A 6-Year Randomized Controlled Trial on Different Implant Designs in Maxillary Overdenture Patients. Clin Implant Dent Relat Res. 2025 Jun;27(3):e70069. doi: 10.1111/cid.70069. PMID 40552788